CLINICAL TRIAL: NCT02595372
Title: Inhibiting Fatty Acid Synthase to Improve Efficacy of Neoadjuvant Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kathy Miller (Other)
Responsible Party: Sponsor-Investigator, Kathy Miller, Professor of Medicine, Ballve' Lantero Scholar, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0555
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Results first posted 2020-06-19 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- High dose omeprazole treatment (Experimental): Patients will be treated with omeprazole 80 mg orally BID beginning 4-7 days prior to chemotherapy and continuing until surgery.
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole

SUMMARY:
In preliminary laboratory science studies, the investigators show that proton pump inhibitors (PPIs) effectively inhibit human fatty acid synthase (FASN) and breast cancer cell survival. A preliminary retrospective study shows that PPI usage in breast cancer patients during chemotherapy significantly improved overall survival. The impact was most striking in patients with triple negative breast cancer (TNBC). Thus, PPIs may be repositioned as safe and effective breast cancer drugs to enhance the effect of chemotherapy.

Many of the hurdles that slow progress from target, to lead compound, to investigational agent, to standard therapy are not barriers for the PPIs. The PPIs are FDA-approved, chronically used, and well tolerated so the investigators can move quickly from the laboratory to a proof of concept clinical trial. Incorporating the PPIs into standard care will require more than the investigators propose here, but the investigators have already plotted the additional steps needed to truly impact patient care. If successful, the data gathered in this proposal will lend support to and guide development of a definitive randomized trial.

DETAILED DESCRIPTION:
Primary Objective

• Estimate the rate of pathologic complete response (pCR) in patients with triple negative breast cancer and FASN expression treated with standard neoadjuvant chemotherapy (NAC) in combination with high dose omeprazole.

Secondary Objectives

* Quantify the number of patients with newly diagnosed TNBC with tumors that express FASN.
* Estimate the rate of pCR in patients with triple negative breast cancer (irrespective of FASN status) treated with standard NAC in combination with high dose omeprazole.
* Describe the safety of incorporating high dose omeprazole with standard NAC.
* Estimate the biologic activity of high dose omeprazole in modulating FASN expression and activity.

This is a single arm Phase II study. Patients should begin therapy within 7 working days of study entry. Patients will be treated with omeprazole 80 mg orally twice a day (BID) beginning 4-7 days prior to chemotherapy and continuing until surgery. After the brief period of omeprazole monotherapy, patients will begin standard neoadjuvant chemotherapy with doxorubicin (60 mg/m2) and cyclophosphamide (600 mg/m2) for 4 cycles followed by paclitaxel (80 mg/m2) weekly x 12. Doxorubicin and cyclophosphamide (AC) may be administered on a classical every 3 week or dose dense every 2 week (with growth factor support) schedule at the treating physician's discretion. Routine incorporation of carboplatin is not recommended, however use of carboplatin (AUC 6 on week 1, 4, 7, and 10) with paclitaxel is allowed at the treating investigator's discretion. Chemotherapy will be adjusted based on toxicity according to standard treatment guidelines. Patients with overt disease progression during AC should move immediately to paclitaxel therapy. Patients with disease progression during paclitaxel should proceed immediately to surgery.

ELIGIBILITY:
Inclusion Criteria

1. Newly diagnosed triple negative breast cancer (TNBC) clinical stage Ic, II, or III

   * ER and PR < 10%
   * HER2 negative based on one of the following:

     * IHC 0 or 1+
     * IHC 2+ and FISH negative
     * IHC 2+ and FISH equivocal and no indication for HER2 targeted therapy based on the treating investigators discretion (i.e., HER2: CEP17 ratio < 2.0 or HER2 total copy number <6)
2. Planned neoadjuvant treatment with anthracycline and taxane containing chemotherapy
3. ≥ 18 years old at the time of informed consent
4. ECOG Performance Status 0-1
5. Ability to provide written informed consent and HIPAA authorization
6. Women of childbearing potential definition must have a negative pregnancy test within 14 days of registration. All women (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) are considered to have childbearing potential unless they meet one of the following criteria:

   * Prior hysterectomy or bilateral oophorectomy;
   * Has not had menses at any time in the preceding 24 consecutive months
7. Adequate organ function for anthracycline and taxane based therapy

   * LVEF > LLN based on cardiac ECHO or MUGA
   * Hgb > 8.5
   * ANC > 1,000
   * Platelets > 100,000
   * Creatinine < 1.5
   * T. bili < 1.3
   * AST < 2.5 x ULN

Exclusion Criteria

1. Use of prescription PPIs within 12 months prior to study entry [Dexlansoprazole (Dexilant), Pantoprazole (Protonix), Rabeprazole (Aciphex), Esomeprazole (Nexium), Lansoprazole (Prevacid), Omeprazole (Prilosec, Zegerid)]
2. Use of OTC PPIs within 6 months prior to study entry [Esomeprazole (Nexium), Lansoprazole (Prevacid), Omeprazole (Prilosec, Zegerid)]
3. Use of Orlistat or any other known FASN inhibitor within 6 months prior to study entry
4. Nursing mothers are excluded
5. Known hypersensitivity to any component of the formulation or substituted benzimidazoles
6. Prior osteoporotic fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Principal Investigator — Professor of Medicine, Ballve' Lantero Scholar
Locations (9):
- United States (9):
  - Georgetown University, Washington D.C., District of Columbia
  - Washington Hospital, Washington D.C., District of Columbia
  - Indiana University Health North Hospital, Carmel, Indiana
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Spring Mill Medical Center, Indianapolis, Indiana
  - Franklin Square Medical Center, Baltimore, Maryland
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Dose Omeprazole Treatment
Started | 42
Completed | 33
Not Completed | 9
Not completed — Adverse Event | 6
Not completed — Physician Decision | 2
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | High Dose Omeprazole Treatment
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 24
  More than one race | 1
  Unknown or Not Reported | 3
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0-Fully active | 36
  1-Restricted in physically strenuous activity | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Pathological Complete Response (pCR) in Patients Who Have Fatty Acid Synthase (FASN) Expression
Description: pCR is defined as no invasive disease in the breast of axilla at the time of definitive surgery. A patient is considered to have FASN expression if the positivity was >= 15% at the baseline or after 4-7 days of Omeprazole monotherapy. FASN expression is evaluated using immunohistochemistry in core biopsy samples. The percent of patients with FASN expression that have pCR will be calculated with an exact 95% confidence interval.
Time Frame: Up to 6 months
Population: Patients who had surgery and positive FASN expression
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High Dose Omeprazole Treatment
Number analyzed (Participants) | 29
percentage of participants | 72.4 [52.8 to 87.3]

2. Secondary Outcome: Percentage of Patients With Pathological Complete Response (pCR) in All Patients
Description: pCR is defined as no invasive disease in the breast or axilla at the time of definitive surgery. The percentage of patients who achieve pCR along with exact 95% confidence intervals were calculated.
Time Frame: Up to 6 months
Population: Patients who received surgery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High Dose Omeprazole Treatment
Number analyzed (Participants) | 39
percentage of participants | 74.4 [57.9 to 87.0]

3. Secondary Outcome: Percent of Patients With FASN Expression
Description: FASN expression was evaluated using immunohistochemistry in core biopsy samples. FASN expression was determined if the positivity was >= 15%. The percent of patients who had FASN expression and the exact 95% confidence intervals were calculated.
Time Frame: up to 1 week
Population: Patients with FASN positivity results at either baseline or after 4-7 days of treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High Dose Omeprazole Treatment
Number analyzed (Participants) | 30
percentage of participants | 93.3 [77.9 to 99.2]

4. Secondary Outcome: FASN Positivity Expression at Baseline and After 4-7 Days of Omeprazole Treatment
Description: The mean and standard deviation of FASN positivity expression determined at baseline and after 4-7 days of Omeprazole treatment. FASN expression is evaluated using immunohistochemistry in core biopsy samples.
Time Frame: baseline and after 4-7 days
Population: Patients with FASN positivity expression at both baseline and after 4-7 days of treatment.
Measure: Mean (Standard Deviation); unit: percentage of positivity
Arm/Group | High Dose Omeprazole Treatment
Number analyzed (Participants) | 24
percentage of positivity
  Baseline | 53.9 (23.6)
  After 4-7 days | 41.7 (30.7)

5. Secondary Outcome: FASN Activity at Baseline and After 4-7 Days of Omeprazole Treatment
Description: The mean and standard deviation of FASN activity determined at baseline and after 4-7 days of Omeprazole treatment. FASN activity was evaluated using immunohistochemistry in core biopsy samples.
Time Frame: baseline and after 4-7 days
Population: Patients with FASN activity evaluated at baseline and after 4-7 days of treatment.
Measure: Mean (Standard Deviation); unit: ng/mg
Arm/Group | High Dose Omeprazole Treatment
Number analyzed (Participants) | 12
ng/mg
  Baseline | 2.1 (1.61)
  After 4-7 days | 1.3 (0.93)

6. Secondary Outcome: Number of Patients With Treatment Related Adverse Events Grade 3 or Above
Description: Number of unique patients who had an Omeprazole treatment related (possible, probable or definite) adverse event with grade >= 3.
Time Frame: up to 8 months
Population: Patients who received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Omeprazole Treatment
Number analyzed (Participants) | 42
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 8 months
Arm/Group | High Dose Omeprazole Treatment
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 5/42
Other Adverse Events (participants affected / at risk) | 37/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Omeprazole Treatment (N=42)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Omeprazole Treatment (N=42)
Anemia (Blood and lymphatic system disorders) | 13
Constipation (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 11
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 7
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 16
Pain (General disorders) | 6
Urinary tract infection (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 10
Neutrophil count decreased (Investigations) | 8
Platelet count decreased (Investigations) | 3
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 9
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 8
Peripheral motor neuropathy (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 16
Anxiety (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 13
Pruritus (Skin and subcutaneous tissue disorders) | 7
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5
Hot flashes (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT02595372/Prot_SAP_000.pdf